CLINICAL TRIAL: NCT02937883
Title: Effects of an Empowerment Intervention for Community-dwelling Persons With Young Onset Dementia and Their Informal Caregivers
Brief Title: Empowerment Intervention for Persons With Young Onset Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 733050607
Record Dates: First submitted 2016-08-01; First posted 2016-10-19 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Dementia; Empowerment
Keywords: Daily Activities
MeSH Terms: conditions — Dementia; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- empowerment intervention (Experimental): Empowerment intervention
  Interventions: Other: Empowerment intervention
- regular care (No Intervention): Regular care, care as usual

INTERVENTIONS:
Other: Empowerment intervention — Empowerment intervention for persons with young onset dementia
  Arms: empowerment intervention

SUMMARY:
The purpose of this study is to evaluate the effects of an empowerment intervention for community-dwelling persons with young onset dementia and their informal caregivers.

DETAILED DESCRIPTION:
This study focuses on the evaluation of an empowerment intervention developed for persons with young onset dementia and their informal caregivers. The empowerment intervention focuses on current capacities, maintenance of autonomy, and increasing the opportunities to feel useful. This pragmatic cluster randomized controlled trial aims to investigate (1) the effectiveness of the intervention concerning participants' well-being, quality of life, and behavioral issues, (2) the effect of the intervention on the informal caregivers' sense of competence and perceived distress, and (3) the impact of the intervention on healthcare costs. Furthermore, the investigators aim to study the feasibility of the intervention to frame an implementation strategy.

Participants in the intervention group will receive the intervention for 5 months. Participants of the control group receive care as usual.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with dementia before the age of 65
* Living at home (community-dwelling)

Exclusion Criteria:

* Dementia is caused by Down's syndrome, Huntington's disease, HIV or alcohol-related dementia.
* Limited contact between the person with dementia and the informal caregiver (<3 times a week)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Changes in self-management abilities | 5 months
  (Self-Management Ability Scale (SMAS))

SECONDARY OUTCOMES:
Changes in quality of life | 5 months
  (Quality of life - Alzheimer Disease scale (QOL-AD))
Changes in neuropsychiatric symptoms Questionnaire | 5 months
  (Neuropsychiatric Inventory (NPI-Q))
Changes in disability | 5 months
  (Interview for Deterioration in Daily living activities in Dementia (IDDD))
Changes in apathy | 5 months
  (abbreviated Apathy Evaluation Scale (AES-10))
Caregiver measures:Competence ( | 5 months
  Short Sense of Competence Questionnaire (SSCQ))
Caregiver measures: Emotional distress | 5 months
  (NPI-Q distress score)

OTHER OUTCOMES:
Analysis of qualitative focus group interviews with participants, caregivers and health care professionals | 5 months
  Qualitative evaluation of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T CM Koopmans, MD, PhD, Principal Investigator — Radboudumc Nijmegen
Locations (1):
- Florence, The Hague, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bielderman A, van Corven CTM, Koopmans RTCM, Leontjevas R, de Vugt ME, Bakker C, Gerritsen DL. Evaluation of the SPAN intervention for people living with young-onset dementia in the community and their family caregivers: a randomized controlled trial. Aging Ment Health. 2024 Jan-Feb;28(2):275-284. doi: 10.1080/13607863.2023.2260335. Epub 2024 Jan 31. PMID 37776001